CLINICAL TRIAL: NCT04088500
Title: A Phase 2, Single-arm Open-label Study of Combination Nivolumab and Ipilimumab Retreatment in Advanced Renal Cell Carcinoma Patients Progressing on Nivolumab Maintenance Therapy After Nivolumab and Ipilimumab Induction
Brief Title: A Study of Combination Nivolumab and Ipilimumab Retreatment in Patients With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-73M
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ipilimumab (combination) (Experimental): Nivolumab + Ipilimumab (combination) Q3W for 4 doses
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specific dose on specific days
  Other Names: Opdivo
Biological: Ipilimumab — Specific dose on specific days

SUMMARY:
The purpose of the study is to assess the effectiveness of re-induction with Nivolumab combined with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

-Participants and Target Disease Characteristics- -

* Confirmed disease progression by RECIST 1.1 criteria on nivolumab maintenance after induction with ipilimumab and nivolumab
* Progress of maintenance treatment of nivolumab by RECIST. Pathology report must be submitted for embedded tissue block or tumor tissue.

Age and Reproduction Sexually active males with WOCBP must agree to instructions for contraception and fetal protection.

WOCBP need to use contraception throughout the study and for 5 months post treatment.

Exclusion Criteria autoimmune disease statement

* Active central nervous system metastases
* Participants with an active autoimmune disease, diabetes mellitus, skin disorders, hyperthyroidism requiring hormone treatments are permitted to enroll.
* Any major surgery 28 days before 1st treatment Concomitant Therapy
* participants that have received a live vaccine within 30 days of treatment.
* use of investigational agent or device with in 28 days before first dosage study treatment.

Physical and Laboratory Test Findings Allergies and Adverse Drug Reaction Age and Reproduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Washington University School of Medicine in St. Louis WUSTL, St Louis, Missouri, United States
- Canada (11):
  - Local Institution, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Atlantic Clinical Cancer Research Unit, Halifax, Nova Scotia
  - Hamilton Health Sciences (HHS) - Juravinski Cancer Centre (JCC), Hamilton, Ontario
  - Toronto Sunnybrook Regional Cancer Ctr, Toronto, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution - 0005, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution - 0006, Sherbrooke, Quebec

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- NIVO 3 + IPI 1: Participants receive ipilimumab 1 mg/kg Q3W combined with nivolumab 3 mg/kg for up to 4 doses followed by nivolumab 480 mg every 4 weeks (Q4W).
Period: Overall Study
Arm/Group | NIVO 3 + IPI 1
Started | 5
Completed | 0
Not Completed | 5
Not completed — Reason unknown | 1
Not completed — Participant withdrew consent | 1
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (11.0)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 2
  >= 65 AND < 75 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is defined as the percentage of participants who achieve a confirmed best response of complete response (CR), partial response (PR), or stable disease (SD) for at least 6 months after first treatment dose per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: From first dose up to approximately 14 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Percentage of participants | 60.0 [14.7 to 94.7]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from first dose to the date of death from any cause. For participants that are alive, their survival time will be censored at the date of last contact ("last known alive date"). OS will be censored for participants at the date of first dose if they were treated but had no follow-up.
Time Frame: From first dose to the date of death from any cause (up to approximately 14 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Months | NA [11.01 to NA] — Insufficient number of participants with events

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) is defined as the percentage of participants who achieve a best response of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose and the date of objectively documented progression criteria or the date of subsequent therapy, whichever occurs first (up to approximately 14 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Percentage of participants | 0.0 [0.0 to 52.2]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) is defined as the time between the date of first documented response (complete response (CR) or partial response (PR)) to the date of the first documented progression, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, or death due to any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to the date of the first documented progression or death due to any cause, whichever occurs first (up to approximately 14 months)
Population: All treated participants with CR or PR
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time between the date of first dose and the first date of documented progression, as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, or death due to any cause, whichever occurs first. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From first dose to the first date of documented progression or death due to any cause, whichever occurs first (up to approximately 14 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Months | NA [4.60 to NA] — Insufficient number of participants with events

6. Secondary Outcome: Time to Objective Response (TTR)
Description: Time to Objective Response (TTR) is defined as the time between the date of the first dose and the first confirmed documented response (complete response (CR) or partial response (PR)) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to the first confirmed documented response (up to approximately 14 months)
Population: All treated participants with CR or PR
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 0

7. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants with any grade adverse events (AEs). An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose and 100 days after lost dose (up to approximately 14 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO 3 + IPI 1
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to approximately 14 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 14 months).
Arm/Group | NIVO 3 + IPI 1
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVO 3 + IPI 1 (N=5)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVO 3 + IPI 1 (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated early, leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04088500/Prot_SAP_000.pdf